CLINICAL TRIAL: NCT06046417
Title: A Randomized, Controlled, Crossover Trial to Assess a Fully Automated, Dual-hormone (Insulin-and-pramlintide) Delivery System Without Carbohydrate Counting in Regulating Glucose Levels in Adults With Type 1 Diabetes.
Brief Title: A Fully Automated Lyumjev and Pramlintide Delivery System for Adults With Type 1 Diabetes
Acronym: FCL
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Michael Tsoukas, Assistant Professor, Endocrinology & Metabolism, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-9373
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: type1diabetes; Diabetes Mellitus, Type 1
Keywords: Pramlintide; fully automated delivery system; artificial pancreas; Insulin; Lyumjev; fully closed loop; adjunctive
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — pramlintide; Insemination, Artificial, Heterologous; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fully automated Lyumjev-and-pramlintide delivery system (8 μg/u) (Experimental): Lyumjev and pramlintide fully automated delivery system with no meal announcement. Ratio of 1 unit of insulin for 8 μg of pramlintide.
  Interventions: Drug: Pramlintide; Drug: Lyumjev; Device: Automated Insulin Delivery (AID) system
- Fully automated Lyumjev-and-pramlintide delivery system (10 μg/u) (Experimental): Lyumjev and pramlintide fully automated delivery system with no meal announcement. Ratio of 1 unit of insulin for 10 μg of pramlintide.
  Interventions: Drug: Pramlintide; Drug: Lyumjev; Device: Automated Insulin Delivery (AID) system
- Hybrid automated Lyumjev-and-placebo delivery system with carbohydrate-matched boluses (Active Comparator): Lyumjev and saline placebo hybrid automated delivery system with meal announcement. Participants must input the carbohydrate content of their meals to inform the insulin bolus doses based on their pre-programmed insulin-to-carbohydrate ratios.
  Interventions: Drug: Lyumjev

INTERVENTIONS:
Drug: Pramlintide — Pramlintide delivered in a basal-bolus manner.
  Arms: Fully automated Lyumjev-and-pramlintide delivery system (10 μg/u); Fully automated Lyumjev-and-pramlintide delivery system (8 μg/u)
Drug: Lyumjev — Lyumjev delivered in a basal-bolus manner.
Device: Automated Insulin Delivery (AID) system — The AID system consists of a set of devices that work inter-connectedly to automate insulin (and pramlintide) delivery in response to an individual's glucose levels. It consists of a (i) Dexcom G6 glucose sensor, (ii) a smartphone-based algorithm, (iii) an insulin YpsoPump, and (iv) a pramlintide/placebo YpsoPump in a dual hormone configuration.
  Arms: Fully automated Lyumjev-and-pramlintide delivery system (10 μg/u); Fully automated Lyumjev-and-pramlintide delivery system (8 μg/u)

SUMMARY:
The aim of this clinical trial is to investigate whether a fully automated Lyumjev-and-pramlintide delivery system improves glycemic outcomes in adults with type 1 diabetes. The main question we aim to answer is whether a Lyumjev-pramlintide fully closed loop system improves time in range compared to a hybrid closed loop system with carbohydrate counting. We also aim to find the optimal insulin to pramlintide ratio for glycemic control in the fully automated system.

In this cross-over study, patients will undergo the following three interventions in a random order:

(i) fully automated Lyumjev insulin-and-pramlintide (8 μg/u) (ii) fully automated Lyumjev insulin-and-pramlintide (10 μg/u) (iii) rapid automated Lyumjev insulin-and-placebo with carbohydrate-matched boluses

For all interventions, participants will be required to wear two Ypsomed pumps programmed by our developed EuGlide system.

DETAILED DESCRIPTION:
The aim of this study is to conduct an outpatient, randomized, crossover clinical trial to compare the glycemic outcomes of a fully automated Lyumjev-pramlintide delivery system to a hybrid automated Lyumjev-placebo delivery system with carbohydrate counting in 26 adults with type 1 diabetes.

Design-

All participants will undergo three interventions in a random order:

(i) Fully automated Lyumjev insulin-pramlintide delivery system. Ratio of 1 unit of inulin for 8μg of pramlintide.

(ii) Fully automated Lyumjev insulin-pramlintide delivery system. Ratio of 1 unit of insulin for 10μg of pramlintide.

(iii) Hybrid automated Lyumjev insulin-placebo delivery system with carbohydrate-matched boluses.

Study drugs-

Lyumjev is a Health Canada insulin for treatment of type 1 diabetes. Participants who do not currently use Lyumjev will be switched to it for the duration of the study.

Pramlintide is an FDA-approved drug used in the treatment of type 1 diabetes. It contributes to regulating glucose levels by delaying gastric emptying, suppressing nutrient-stimulated glucagon secretion and increasing satiety. It is not approved for commercial use by Health Canada, but has been approved for the purpose of the study.

Study Devices-

For the duration of the study, participants will use a Dexcom G6 Continuous Glucose Monitor (GCM), two YpsoPumps (for insulin and pramlintide) as well as a study smartphone with the Euglide application installed. The automated insulin delivery (AID) system will integrate these sets of devices to automate insulin (and pramlintide) delivery in response to an individual's glucose levels.

Treatment Period-

Each intervention will last three weeks and be preceded by a 5-day at-home run-in period. After both the second and third interventions, there will be a 14-45 day washout period. Participants will be followed-up with remotely on days 2 (+/-1) and 5 of each run-in and on days 2(+/-1), 3(+/-1) and 7(+/-2) of each intervention. Remote contact can be performed via phone, email, text message or another reasonable communication channel. After each intervention, participants will be interviewed and asked to complete questionnaires assessing diabetes control and quality of life. Participants will need approximately 15-30 weeks to complete the study.

The study will enroll up to 4 pilot participants, as well as 26 main study participants who meet the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 18 years of age.
* A clinical diagnosis of type 1 diabetes for at least 12 months. The diagnosis of type 1 diabetes relies on the investigator's judgment; C peptide level and antibody determinations are unnecessary.
* Using insulin pump therapy for at least three months.
* Individuals of childbearing potential using an effective birth-control method. An individual of childbearing potential must agree to use a highly effective method of birth control.

Exclusion Criteria:

* Current or recent use of antihyperglycemic agents other than insulin (≤ 2-week use of sodium-glucose cotransporter-2 inhibitor (SGLT2I), Metformin, etc.; ≤ 1-month for glucagon-like peptide-1 receptor agonists (GLP1-RA)).
* Current use of glucocorticoid medication (except low, stable doses and inhaled steroids).
* Individuals with confirmed gastroparesis.
* Use of medication that alters gastrointestinal motility (ex: domperidone).
* Use of hydroxyurea.
* Planned or ongoing pregnancy.
* Breastfeeding individuals.
* Severe hypoglycemia requiring hospitalization in the past month. Severe hypoglycemia is defined as requiring the assistance of another person, due to altered consciousness, to administer carbohydrates, glucagon, or other resuscitative actions.
* Diabetic ketoacidosis episode in the past month.
* Clinically significant nephropathy, neuropathy, or retinopathy as judged by the investigator.
* Recent (< 6 months) acute macrovascular event, e.g., acute coronary syndrome.
* Other serious medical illnesses which are likely to interfere with study participation or the ability to complete the trial by the investigator's judgment.
* Known hypersensitivity to the study drugs or their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of time of glucose levels spent in the target range (3.9-10.0 mmol/L). | 18 days

SECONDARY OUTCOMES:
Percentage of time of glucose levels spent between 3.9-7.8 mmol/L. | 18 days
Percentage of time of glucose levels spent between 3.0-3.9 mmol/L. | 18 days
Percentage of time of glucose levels spent between 10.0-13.9 mmol/L. | 18 days
Mean glucose levels. | 18 days
Standard deviation of glucose levels. | 18 days
Coefficient of variance of glucose levels. | 18 days
Total pramlintide delivery (overall, basal, and bolus). | 18 days
Total insulin delivery (overall, basal, and bolus). | 18 days
Mean score on the Type 1 Diabetes Distress Scale (T1DDS) excluding the physician subscale. | 18 days
  A scale from 1-6 indicating overall diabetes distress. Higher scores indicate higher levels of diabetes distress. Any total subscale score of >2.0 is considered clinically significant.
Mean score on the Hypoglycemia Fear Survey - II (Worry Subscale) (HSF2). | 18 days
  A scale from 1-5 with higher scores indicating a greater fear of hypoglycemia.
Mean score on the INSPIRE questionnaire for adults (INSPIRE). | 18 days
  A scale from 1-5 with higher scores reflecting more favorable opinions about using Automated Insulin Delivery (AID).
Mean score on selected items from The Diabetes Bowel Symptoms Questionnaire (DBSQ). | 18 days
  A 1-5 scale with higher values reflecting a greater quantity and severity of diabetes bowel symptoms.
Mean score on a Treatment Satisfaction Questionnaire (TSQ) taken from Marrero et al. | 18 days
  A 1-6 scale with higher values indicating more satisfaction with treatment.
Thematic interview analysis | 18 days
  Semi-structured interviews will be carried out after every intervention. We will analyze their qualitative content.

OTHER OUTCOMES:
Safety Endpoints | 18 days
  Number of adverse events, including gastrointestinal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tsoukas, M.D., Principal Investigator — Research Institute of the McGill University Health Center; Ahmad Haidar, Ph.D., Study Chair — Research Institute of the McGill University Health Center; Laurent Legault, M.D., Study Chair — Montreal's Children's Hospital Division of Endocrinology; Michael Vallis, Ph.D., Study Chair — Dalhousie University Psychologist; Natasha Garfield, M.D., Study Chair — Royal Victoria Hospital Division of Endocrinology; Melissa-Rosina Pasqua, M.D., Study Chair — Research Institute of the McGill University Health Center
Locations (1):
- Research Institute of the McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The raw data (that is, insulin delivery, glucose levels and individual participant data) and informed consent form will be shared by the corresponding author, for academic purposes, subject to a material transfer agreement and approval of the McGill University Health Center's Research Ethics Board. All data shared will be de-identified. Raw data will be shared for non-commercial use upon reasonable request and a material transfer agreement.
Supporting Information: ICF